CLINICAL TRIAL: NCT06171464
Title: Prognostic Value of Pre-therapy 18F-FDG PET/CT for the Outcome of 18 FDG PET-guided SIB-IMRT in Patients With Head and Neck Cancer
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Chiti Arturo, Professor in Diagnostic Imaging and Radiotherapy Faculty of Medicine and Surgery, Vita-Salute San Raffaele University Director, Department of Nuclear Medicine, IRCCS Ospedale San Raffaele, IRCCS San Raffaele
Other Study IDs: PETCT-PRERT-HNC
Record Dates: First submitted 2023-12-04; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Head and neck cancer is the fifth most common cancer and represents 5% in the world.

Selecting patients for the most appropriate treatment remains difficult. Approximately 60-65% of patients undergo surgery followed or not by radiotherapy. Patients with early stage disease (I-II) are treated with one treatment modality (surgery or radiotherapy), while patients with more advanced stage disease (III-IV) receive multimodal treatment (surgery together with associated radiotherapy or less to chemotherapy). PET/CT plays a fundamental role in the management of head and neck cancer patients. This investigation is indicated for staging, especially in patients with disease in advanced stages, for evaluating the response to therapy and for looking for recurrences as it is more accurate in distinguishing scar tissue from neoplasm. The objective of this retrospective study is to evaluate the prognostic value of PET/CT in predicting the outcome of patients undergoing SlB-IMRT/intensity modulated radiotherapy). The study proposed here involves the retrospective recruitment of patients who have performed a PET/CT investigation with 18F-FDG (fluorodeoxyglucose) at the U.O. of HSR Nuclear Medicine in the staging and treatment planning phase, between 2005 and 2011. The inclusion condition of the patients was their PET/CT evaluation (planning and treatment) using the "DSTE" PET/CT system installed at the U.O. of Nuclear Medicine HSR on which, in the presence of homogeneous lesions. a particular correction technique is applicable, developed and validated previously by the research group, which allows possible metabolic markers to be extracted from the lesions in a quantitatively accurate way.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from head and neck cancer;
* patients who underwent PET-CT with 18F-FDG.

Exclusion Criteria:

* patients <18 years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients suffering from head and neck cancer who performed a PET-CT investigation with 18F-FDG for treatment planning with Intensity modulated Radiotherapy with integrated simultaneous boost (IMRT-SIB).
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2013-02-21 (Actual); Primary Completion 2013-12-01 (Actual); Study Completion 2013-12-01 (Actual)

PRIMARY OUTCOMES:
PET-CT investigation with 18F-FDG for staging patients with head and neck cancer. | 1 year
  Patients underwent 18 F-FDG PET-CT during staging and treatment planning. They subsequently underwent Intensity Modulated Radiotherapy (IMRT) with a simultaneous boost (SIB) on a region highlighted by PET-CT as metabolically active.